CLINICAL TRIAL: NCT05582993
Title: A Phase 3, Prospective, Open-label, Uncontrolled, Multicenter Study on Efficacy and Safety of Prophylaxis With Vonicog Alfa (rVWF) in Children Diagnosed With Severe Von Willebrand Disease
Brief Title: A Study of Vonicog Alfa (rVWF) in Children With Severe Von Willebrand Disease (vWD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-577-3001; 2023-509877-22-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-14; First posted 2022-10-17 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Von Willebrand Disease (VWD)
MeSH Terms: conditions — von Willebrand Diseases | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Participants With Age >=12 to <18 years (Experimental): Participants with age greater than or equal to (>=) 12 to less than (<) 18 years who have received on-demand (OD) therapy or prophylactic treatment with a pdVWF product will receive vonicog alfa (rVWF) with an initial dose selected within the range of 40 to 60 international units per kilogram (IU/kg) vonicog alfa (rVWF), intravenous infusions, twice-weekly for 12 months. Participants may receive vonicog alfa (rVWF) with or without ADVATE intravenous infusions, when indicated (as deemed necessary for breakthrough bleeding episode treatment and perioperative bleeding management).
  Interventions: Biological: Vonicog Alfa; Biological: ADVATE
- Cohort 2: Participants With Age >=6 to <12 years (Experimental): Participants with age >=6 to <12 years who have received OD therapy of VWF product or prophylactic treatment with a pdVWF product will receive vonicog alfa (rVWF) with an initial dose selected within the range of 40 to 60 IU/kg vonicog alfa (rVWF), intravenous infusions, twice-weekly for 12 months. Participants may receive vonicog alfa (rVWF) with or without ADVATE intravenous infusions, when indicated (as deemed necessary for breakthrough bleeding episode treatment and perioperative bleeding management).
  Interventions: Biological: Vonicog Alfa; Biological: ADVATE
- Cohort 3: Participants With Age <6 years (Experimental): Participants with age <6 years who have received OD therapy of VWF product or prophylactic treatment with a pdVWF product will receive vonicog alfa (rVWF) with an initial dose selected within the range of 40 to 60 IU/kg vonicog alfa (rVWF), intravenous infusions, twice-weekly for 12 months. Participants may receive vonicog alfa (rVWF) with or without ADVATE intravenous infusions, when indicated (as deemed necessary for breakthrough bleeding episode treatment and perioperative bleeding management).
  Interventions: Biological: Vonicog Alfa; Biological: ADVATE

INTERVENTIONS:
Biological: Vonicog Alfa — Vonicog Alfa administered by intravenous injection.
  Other Names: TAK-577; Recombinant von Willebrand Factor (rVWF); Vonvendi-Veyvondi
Biological: ADVATE — ADVATE administered by intravenous injection.
  Other Names: Recombinant Factor VIII (rFVIII); Octocog Alfa

SUMMARY:
The main aim of the study is to evaluate the effectiveness of prophylaxis with vonicog alfa (recombinant von Willebrand factor [rVWF]) in children. This study will enroll those participants who have been previously treated with VWF product or with a plasma-derived VWF (pdVWF) product. In this study, participants will be treated with vonicog alfa (rVWF) for 12 months.

During the study, participants will visit the study clinic 5 times after treatment initiation.

ELIGIBILITY:
1. The participant has a documented diagnosis of severe VWD (baseline von Willebrand factor ristocetin cofactor activity [VWF:RCo] <20 international units per deciliter [IU/dL]) with a history of replacement therapy with VWF concentrate required to control bleeding and a diagnosis of VWD type 1, type 2 (2A, 2B, 2M, 2N), or type 3. Diagnosis is confirmed, as applicable, by genetic testing and/or by multimer analysis, which may be documented in participant's history or at screening.
2. The participant is <18 years of age at the time of screening.
3. Prescreening treatment requirements:

   1. The participant has been receiving OD therapy with VWF products for at least 12 months (for participants >=2 years of age) prior to screening, has experienced at least 1 VWF-treated bleeding event during (excluding menorrhagia/heavy menstrual bleeding [HMB], as applicable) in the last 12 months, and prophylactic treatment is recommended by the investigator (Prior OD participants); or
   2. The participant has been receiving prophylactic treatment with pdVWF products for at least 12 months prior to screening (for participants >=2 years of age) and switching to prophylaxis with vonicog alfa (rVWF) is recommended by the investigator (Switch participants).
   3. For participants <2 years of age, the required duration for prior OD therapy with VWF products or for prior prophylactic treatment with pdVWF products is at least 6 months. Prior OD participants <2 years of age should have experienced at least 1 VWF-treated bleeding event during the last 6 months based on medical records and be recommended to receive prophylactic treatment by the investigator.
4. For participants >=2 years of age, the participant has available records that reliably evaluate type, frequency, severity, and treatment of BEs for at least 12 months preceding enrollment. For participants <2 years of age, the participant has available records that reliably evaluate type, frequency, severity and treatment of BEs for at least 6 months preceding enrollment.
5. If >=12 years old at the time of screening, the participant has a body mass index (BMI) >=15 but <40 kilogram per square meter (kg/m^2). If >=2 to <12 years old at the time of screening, the participant has a BMI of >=5th and <95th percentile (per Centers for Disease Control and Prevention [CDC] clinical charts). For younger participants who are <2 years old, the "weight-for-age" clinical charts (5th to 95th percentile) provided by the CDC should be utilized to ensure the participant has a body weight of >=5th and <95th percentile based on gender (for clinical charts provided by CDC, refer to: https://www.cdc.gov/growthcharts/clinical_charts.htm).
6. Female participants of childbearing potential (that is, had onset of menses/reached puberty) must have a negative blood/urine pregnancy test result at screening and agree to employ highly effective birth control measures for the duration of their participation in the study.
7. The participant has voluntarily provided assent (if appropriate) and the legally authorized representative(s) has provided informed consent.
8. The participant and/or legally authorized representative is willing and able to comply with the requirements of the protocol, which should also be confirmed based on a prescreening evaluation held between the investigator and the sponsor to ensure no eminent risk is present that could challenge the participant's compliance with the study requirements.

Exclusion Criteria:

1. The participant has been diagnosed with pseudo VWD or another hereditary or acquired coagulation disorder other than VWD (example, qualitative and quantitative platelet disorders or elevated prothrombin time/international normalized ratio 1.4).
2. The participant has a history or presence of a VWF inhibitor at screening.
3. The participant has a history or presence of an factor VIII (FVIII) inhibitor with a titer >=0.6 Bethesda units per milliliter (/mL).
4. The participant has a known hypersensitivity to any of the components of the study drugs, such as mouse or hamster proteins.
5. The participant has a medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis, mild asthma, food allergies, or animal allergies.
6. The participant has a medical history of a thromboembolic event.
7. The participant is human immunodeficiency virus (HIV)-positive with an absolute helper T cell (CD4) count <200 per cubic millimeter or microliter (/mm^3).
8. The participant has been diagnosed with significant liver disease per the investigator's medical assessment of the participant's current condition or medical history or as evidenced by, but not limited to, any of the following: serum alanine aminotransferase (ALT) greater than 5 times the upper limit of normal (ULN), hypoalbuminemia, portal vein hypertension (example, presence of otherwise unexplained splenomegaly, history of esophageal varices), or liver cirrhosis classified as Child-Pugh class B or C.
9. The participant has been diagnosed with renal disease, with a serum creatinine level >=2.5 milligram per deciliter (mg/dL).
10. The participant has a platelet count <100,000/mL at screening (because participants with type 2B VWD are considered eligible for this study, for participants with type 2B VWD, platelet count[s] at screening will be evaluated in consultation with the sponsor, taking into consideration historical trends in platelet counts and the investigator's medical assessment of the participants condition).
11. The participant has been treated with an immunomodulatory drug, excluding topical treatment (example, ointments, nasal sprays), within 30 days prior to signing the informed consent (or assent, if appropriate).
12. The participant is pregnant or lactating at the time of enrollment.
13. The participant has cervical or uterine conditions causing menorrhagia or metrorrhagia (including infection, dysplasia).
14. The participant has participated in another clinical study involving another IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
15. The participant has not received OD or prophylactic treatment with a VWF product prior to this study.
16. The participant has a progressive fatal disease and/or life expectancy of less than 15 months.
17. The participant is unable to complete screening procedures and/or comply with the requirements of the protocol in the opinion of the investigator, based on the joint prescreening evaluation held between the investigator and the sponsor.
18. The participant has a mental condition rendering him/her unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude.
19. The participant is member of the study team or in a dependent relationship with one of the study team members, which includes close relatives (that is, children, partner/spouse, siblings, and parents) as well as employees.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2030-04-11 (Estimated); Study Completion 2030-04-11 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) for Spontaneous or Traumatic Bleeding Episodes as Assessed by Investigator During Prophylactic Treatment With Vonicog Alfa (rVWF) | 12 months
  ABR during the study compared to historical ABR for each participant for both spontaneous and traumatic bleeding episodes as classified by the investigator during prophylactic treatment with vonicog alfa (rVWF) will be reported.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 12 months
  Number of participants with TEAEs and SAEs will be reported.
Number of Participants With TEAEs by Severity | 12 months
  Number of participants with severity of TEAE will be reported.
Number of Participants With TEAEs and SAEs by Causality | 12 months
  Number of participants with causality related TEAEs and SAEs will be reported.
Number of Participants With Thromboembolic Events, Hypersensitivity Reactions and Infusion-Related Reactions (IRR) | 12 months
  Number of participants with thromboembolic events, hypersensitivity reactions and IRR will be reported.
Number of Participants Who Develop Neutralizing Antibodies to VWF and Factor VIII (FVIII) | 12 months
  Number of participants who develop neutralizing antibodies to VWF and FVIII will be reported.
Number of Participants Who Develop Binding Antibodies to VWF and FVIII | 12 months
  Number of participants who develop total binding antibodies to VWF and FVIII will be reported.
Number of Participants With Clinically Significant Change From Baseline Values in Vital Sign Parameters | 12 months
  Number of participants with clinically significant change from baseline values in vital sign parameters per investigator assessment will be reported.
Number of Participants With Clinically Significant Change From Baseline Values in Laboratory Parameters | 12 months
  Number of participants with clinically significant change from baseline values in laboratory parameters per investigator assessment will be reported.
Number of Participants With Categorized ABR | 12 months
  ABR categorized as 0, 0-2, 2-5, or >5 bleeding episodes during vonicog alfa (rVWF) prophylaxis. Number of participants with categorized ABR will be reported.
Number of Participants Previously Receiving On-demand Treatment who will Achieve ABR Percent Reduction Success | 12 months
  ABR percent reduction success is defined as at least 25% reduction of ABR during vonicog alfa (rVWF) prophylaxis relative to the participant's own historical ABR during OD treatment prior to enrollment in this study. Number of participants previously receiving on-demand treatment who will achieve ABR percent reduction success will be reported.
Number of pdVWF Switch Participants With Spontaneous ABR Preservation Success | 12 months
  ABR preservation success is defined as achieving an ABR for spontaneous bleeding episodes during vonicog alfa (rVWF) prophylaxis that is no greater than the participant's own historical ABR during prophylactic treatment with pdVWF prior to enrollment in this study. Number of pdVWF switch participants with spontaneous ABR preservation success will be reported.
Number of Spontaneous ABR Historically and While on Prophylactic Treatment With Vonicog Alfa (rVWF) by Location of Bleeding | 12 months
  Number of spontaneous ABR historically and while on prophylactic treatment with vonicog alfa (rVWF) by location of bleeding will be reported.
ABR for Bleeding Episodes by Bleeding Cause Historically and While on Prophylactic Treatment With Vonicog Alfa (rVWF) | 12 months
  ABR for bleeding episodes by bleeding cause historically and while on prophylactic treatment with vonicog alfa (rVWF) will be reported.
Total Number of Infusions Administered Per Week During Prophylactic Treatment With Vonicog Alfa (rVWF) | 12 months
  Total number of infusions administered per week during prophylactic treatment with vonicog alfa (rVWF) will be reported.
Average Number of Infusions Per Week During Prophylactic Treatment With Vonicog Alfa (rVWF) | 12 months
  Average number of infusions per week during prophylactic treatment with vonicog alfa (rVWF) will be reported.
Total Weight Adjusted Consumption of Vonicog Alfa (rVWF) Per Month During Prophylactic Treatment | 12 months
  Total weight adjusted consumption of vonicog alfa (rVWF) per month during prophylactic treatment will be reported.
Overall Hemostatic Efficacy Rating of Breakthrough Bleed Treatment at Resolution of the Bleeding Episode | 12 months
  Overall hemostatic efficacy rating of breakthrough bleed treatment at resolution of the bleeding episode will be reported.
Number of Infusions of rVWF and ADVATE (rFVIII, octocog alfa) per Bleeding Episode | 12 months
  Number of infusions of vonicog alfa (rVWF) and ADVATE per bleeding episode will be reported.
Weight-adjusted Consumption of Vonicog Alfa (rVWF) and ADVATE per Bleeding Episode | 12 months
  Weight-adjusted consumption of vonicog alfa (rVWF) and ADVATE per bleeding episode will be reported.
Plasma Level of Vonicog Alfa (rVWF) based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Plasma level of vonicog alfa (rVWF) based on VWF:Rco will be reported.
Plasma Level of Vonicog Alfa (rVWF) based on Von Willebrand Factor Antigen (VWF:Ag) | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Plasma level of vonicog alfa (rVWF) based on VWF:Ag will be reported.
Plasma Level of Vonicog alfa (rVWF) based on Von Willebrand Factor Collagen Binding (VWF:CB) | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Plasma level of vonicog alfa (rVWF) based on VWF:CB will be reported.
Plasma Level of Vonicog alfa (rVWF) based on Von Willebrand Factor Glycoprotein 1b Binding (VWF:GP1bM) | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Plasma level of vonicog alfa (rVWF) based on VWF:GP1bM will be reported.
Plasma Level of Factor VIII Clotting (FVIII:C) | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Plasma level of FVIII:C will be reported.
Incremental Recovery Based on VWF:Rco | 12 months
  Incremental recovery based on VWF:Rco will be reported.
Incremental Recovery Based on VWF:Ag | 12 months
  Incremental recovery based on VWF:Ag will be reported.
Incremental Recovery Based on VWF:CB | 12 months
  Incremental recovery based on VWF:CB will be reported.
Incremental Recovery Based on VWF:GP1bM | 12 months
  Incremental recovery based on VWF:GP1bM will be reported.
Ratio of Area Under the Plasma Level Versus Time Curve From Time 0 to End of the Partial Dosing Interval (AUC0- Tau;ss) and Area Under the Level Versus Time Curve From 0 to 96 Hours (AUC0-96; ss) for VWF:Rco | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Ratio of AUC0- Tau;ss/AUC0-96; ss for VWF:Rco will be reported.
Terminal Half-life (T1/2) for VWF:Rco | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  TT1/2 based on VWF:Rco will be reported.
Maximum Plasma Level During the Partial Dosing Interval at Steady State (Cmax;ss) for VWF:Rco | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Cmax;ss for VWF:Rco will be reported.
Minimum Time to Reach the Maximum Plasma Level at Steady State (Tmax;ss) for VWF:Rco | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Tmax;ss for VWF:Rco will be reported.
Volume of Distribution at Steady State (Vss) for VWF:Rco | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Vss for VWF:Rco will be reported.
Clearance (CL) for VWF:Rco | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  CL for VWF:Rco will be reported.
Maximum Plasma Level During the Partial Dosing Interval at Steady State (Cmax;ss) for FVIII:C | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Cmax;ss for FVIII:C will be reported.
Minimum Time to Reach the Maximum Plasma Level at Steady State (Tmax;ss) for FVIII:C | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Tmax;ss for FVIII:C will be reported.
Ratio of Area Under the Plasma Level Versus Time Curve From Time 0 to End of the Partial Dosing Interval (AUC0- Tau;ss) and Area Under the Level Versus Time Curve From 0 to 96 Hours (AUC0-96; ss) for FVIII:C | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  Ratio of AUC0- Tau;ss and AUC0-96; ss for FVIII:C will be reported.
Area Under the Level Versus Time Curve From 0 to 96 Hours (AUC0-96; ss) for FVIII:C | Within 30 minutes pre-infusion and at multiple timepoints (up to 96 hours) post-infusion
  AUC0-96; ss for FVIII:C will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Riley Hospital for Children Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics PARENT, Iowa City, Iowa
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Children's Health Care d/b/a Children's Minnesota, Minneapolis, Minnesota
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York - Presbyterian/Weill Cornell Medical Center, New York, New York
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
- France (2):
  - Hemostase Clinique - Institut Cœur-Poumons (4eme étage aile est) Bureau 419, Lille
  - Hopital Edouard Herriot - CHU Lyon, Lyon
- Children's Health Ireland, Dublin, Ireland
- Italy (2):
  - Azienda Ospedaliera Pediatrica Santobono Pausillipon, Napoli
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Turin (Torino)
- Nara Medical University Hospital, Kashihara, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/b48da778c86b4f5a?idFilter=%5B%22TAK-577-3001%22%5D